CLINICAL TRIAL: NCT02525003
Title: Work Package 5: The Potential Advantages and Limitations of Use of Novel Food-based Solutions for Prevention of Vitamin D Deficiency. Food-based Solutions for Optimal Vitamin D Nutrition and Health Through the Life Cycle (ODIN)
Brief Title: The BreaD Study - Bio-availability of D2 Vitamin Present in Bread
Acronym: BreaD_ODIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University College Cork (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Christel Lamberg-Allardt, Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HelsinkiUni
Record Dates: First submitted 2015-08-10; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Serum 25-hydroxyvitamin D Concentrations (25OHD)
Keywords: vitamin D; Serum 25-hydroxyvitamin D; vitamin D2; UV-irradiated yeast; serum 25-hydroxyvitamin D3; serum 25-hydroxyvitamin D2; randomized controlled trial; vitamin D3; bioavailability
MeSH Terms: interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: placebo (Placebo Comparator): Group 1: daily dose of regular bread (87 g/d) and placebo pill (0 µg of vitamin D/d) for 8 weeks
- Group 2: Vitamin D2 supplement (Experimental): Group 2: daily dose of regular bread (87 g/d) and D2 supplement (25 µg of vitamin D2/d.) for 8 weeks
  Interventions: Dietary Supplement: Vitamin D2
- Group 3: Vitamin D3 supplement (Experimental): Group 3: daily dose of regular bread (87 g/d) and D3 supplement (25 µg of vitamin D3/d.) for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Group 4: Vitamin D2-fortified bread (Experimental): Group 4: D2 fortified bread containing 25 µg of vitamin D2/d (bread dose 87g/d) and placebo pill for 8 weeks
  Interventions: Other: Vitamin D2 fortified bread

INTERVENTIONS:
Dietary Supplement: Vitamin D2 — Experimental group 2: daily vitamin D2 supplement 25ug/d for 8 weeks
  Arms: Group 2: Vitamin D2 supplement
Dietary Supplement: Vitamin D3 — Experimental group 3: daily vitamin D3 supplement 25ug/d for 8 weeks
  Arms: Group 3: Vitamin D3 supplement
Other: Vitamin D2 fortified bread — Experimental group 4: vitamin D2 fortified bread containing 25 µg of vitamin D2/d (bread dose 87g/d) and placebo pill for 8 weeks
  Arms: Group 4: Vitamin D2-fortified bread

SUMMARY:
Vitamin D3 is synthesized in skin exposed to ultraviolet-B-irradiation of sunlight. However, in Northern Europe, including Finland, exposure to sunlight is limited or non-existent in winter. Between November and March, dietary or supplementary vitamin D intake is essential to maintain adequate serum 25-hydroxyvitamin D (S-25(OH)D) concentrations. There are only a few natural dietary sources of vitamin D. Fish and egg yolks contain significant amounts of vitamin D3 (cholecalciferol), and some wild mushrooms are a source of vitamin D2 (ergocalciferol). Thus, vitamin D fortification of certain foods has been accepted as one strategy to improve vitamin D status of these populations. Vitamin D3 is currently mostly used in fortified products in Europe, although the production of plant-derived vitamin D2 would be more cost-effective. Data on the impact of food-derived vitamin D2 on S-25(OH)D3 are limited. An important consideration is whether food-based sources of vitamin D2 are effective in raising S-25(OH)D or whether they have a negative impact on S-25(OH)D3. The investigators investigated the bioavailability of vitamin D2 from UVB-radiated baking yeast in bread in terms of efficacy of raising total S-25(OH)D) as well its possible effects on S-25(OH)D2, S-25(OH)D3, serum parathyroid hormone (S-PTH) and serum calcium concentrations compared with D2 and D3 supplementation in a randomized placebo-controlled trial in young healthy females during winter in Finland.

ELIGIBILITY:
Inclusion Criteria:

* good general health (no continuous medication),
* Caucasian origin,
* body mass index (BMI) <30 kg/m2
* age 20-40 years

Exclusion Criteria:

* diagnosed celiac disease or cereal allergy
* a vacation in a sunny place during the study or within the preceding 2 months
* regular use of vitamin D supplements >15 µg/d
* pregnancy or breastfeeding during the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Serum total 25-hydroxyvitamin D (25(OH)D) | Change from baseline in total 25(OH)D concentration at 4 and 8 weeks
  The effect of vitamin D (as form of D3, D2 or D2-fortified bread )supplementation on the serum 25(OH)D concentration

SECONDARY OUTCOMES:
Serum parathyroid hormone (PTH) concentration | Change from baseline in serum PTH concentration at 4 and 8 weeks
  The effect of vitamin D (as form of D3, D2 or D2-fortified bread )supplementation on the serum PTH concentration
Serum calcium concentration | Change from baseline in serum calcium concentration at 4 and 8 weeks
  The effect of vitamin D (as form of D3, D2 or D2-fortified bread )supplementation on the serum calcium concentration
Serum 25-hydroxyvitamin D2 (25(OH)D2) | Change from baseline in 25(OH)D2 concentration at 4 and 8 weeks
  The effect of vitamin D (as form of D3, D2 or D2-fortified bread )supplementation on the serum 25(OH)D2 concentration
Serum 25-hydroxyvitamin D3 (25(OH)D3) | Change from baseline in 25(OH)D3 concentration at 4 and 8 weeks
  The effect of vitamin D (as form of D3, D2 or D2-fortified bread )supplementation on the serum 25(OH)D3 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Christel Lamberg-Allardt, Study Director — University of Helsinki
Locations (1):
- Department of Food and Environmental Sciences, University of Helsinki, Helsinki, Finland